CLINICAL TRIAL: NCT02228148
Title: Comparison of Fitting Methods Using Cochlear Clinical Care Innovation
Brief Title: Comparison of the New Fitting Method Cochlear Nucleus Fitting Software (NFS) With the Established Fitting Method Cochlear Nucleus Custom SoundTM Suite (CSS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: numerics data GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEL5332
Record Dates: First submitted 2014-08-27; First posted 2014-08-28 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
Keywords: Post linguistically deafness, severe to profound deafness
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NFS (Experimental): Cochlear Nucleus Fitting Software
  Interventions: Device: NFS
- CSS (Active Comparator): Cochlear Nucleus Custom SoundTM Suite
  Interventions: Device: CSS

INTERVENTIONS:
Device: NFS — Cochlear Nucleus Fitting Software
  Arms: NFS
Device: CSS — Cochlear Nucleus Custom SoundTM Suite
  Arms: CSS

SUMMARY:
The purpose of this study is to evaluate if the new and simplified fitting method with Cochlear Nucleus Fitting Software (a major component of a suite of tools which form the Clinical Care Innovation) provides Cochlear Implants Recipients with the same hearing outcome as the current and established clinical fitting method with Cochlear Nucleus Custom SoundTM Suite. The Clinical Care Innovation method reduces fitting to simple volume, bass and trebles adjustments, operations which are familiar to anyone who has used an audio player.

ELIGIBILITY:
Inclusion Criteria:

* Newly implanted subjects with available Nucleus Cochlear Implants compatible with CP900 series sound processors (excluding Cochlear Nucleus Hybrid)
* Post linguistically deafened adults (≥ 18 years)
* Unilaterally implanted
* ≤ 15 years of severe to profound deafness prior to implantation
* Subjects who are capable and willing to participate in speech perception tests in local language
* Subjects who are able to provide feedback in form of a written questionnaire (e.g. Speech Spatial Hearing Qualities questionnaire)
* Subjects willing to give their consent to the study

Exclusion Criteria:

* Additional handicaps that would prevent participation in evaluations (e.g. visual impairment, blindness)
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure/fitting method
* Bilateral implantation
* Hybrid-L (not supported by Nucleus Fitting Software)
* Subjects who already have hearing experience with a Cochlear Implant (e.g. reimplantation, contralateral Cochlear Implant)
* Subjects with single-sided deafness
* Known cochlea malformations
* Subjects who lost their hearing due to meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via aided hearing thresholds | 3 months after implantation
  Adaptive Oldenburg Sentence Test in noise with speech at 65 dB (if the subject's understanding with Oldenburg Sentence Test in quiet is ≥ 70%).
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via aided hearing thresholds | 6 months after implantation
  Adaptive Oldenburg Sentence Test in noise with speech at 65 dB (if the subject's understanding with Oldenburg Sentence Test in quiet is ≥ 70%).
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via aided hearing thresholds | 9 months after implantation
  Adaptive Oldenburg Sentence Test in noise with speech at 65 dB (if the subject's understanding with Oldenburg Sentence Test in quiet is ≥ 70%).
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via aided hearing thresholds | 12 months after implantation
  Adaptive Oldenburg Sentence Test in noise with speech at 65 dB (if the subject's understanding with Oldenburg Sentence Test in quiet is ≥ 70%).
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via aided hearing thresholds | 15 months after implantation
  Adaptive Oldenburg Sentence Test in noise with speech at 65 dB (if the subject's understanding with Oldenburg Sentence Test in quiet is ≥ 70%).
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via speech performance tests | 3 months after implantation
  Freiburg Monosyllables and Oldenburg Sentence Test in quiet at 65 dB.
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via speech performance tests | 6 months after implantation
  Freiburg Monosyllables and Oldenburg Sentence Test in quiet at 65 dB.
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via speech performance tests | 9 months after implantation
  Freiburg Monosyllables and Oldenburg Sentence Test in quiet at 65 dB.
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via speech performance tests | 12 months after implantation
  Freiburg Monosyllables and Oldenburg Sentence Test in quiet at 65 dB.
Speech perception performance in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via speech performance tests | 15 months after implantation
  Freiburg Monosyllables and Oldenburg Sentence Test in quiet at 65 dB.

SECONDARY OUTCOMES:
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | before first fitting post-implantation (1 day)
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | 3 months after implantation
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | 6 months after implantation
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | 9 months after implantation
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | 12 months after implantation
Hearing disability score in subjects fitted with Nucleus Fitting Software and subjects fitted with Nucleus Custom SoundTM Suite assessed via the Speech Spatial Hearing Qualities questionnaire (without spatial part) | 15 months after implantation
Subject preference for fittings performed with Nucleus Fitting Software and fittings with Nucleus Custom SoundTM Suite assessed via a subject comfort questionnaire | after each fitting (4 weeks after implantation)
Subject preference for fittings performed with Nucleus Fitting Software and fittings with Nucleus Custom SoundTM Suite assessed via a subject comfort questionnaire | after each fitting (3 months after implantation)
Subject preference for fittings performed with Nucleus Fitting Software and fittings with Nucleus Custom SoundTM Suite assessed via a subject comfort questionnaire | after each fitting (6 months after implantation)
Subject preference for fittings performed with Nucleus Fitting Software and fittings with Nucleus Custom SoundTM Suite assessed via a subject comfort questionnaire | after each fitting (9 months after implantation)
Subject preference for fittings performed with Nucleus Fitting Software and fittings with Nucleus Custom SoundTM Suite assessed via a subject comfort questionnaire | after each fitting (12 months after implantation)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, PhD, Study Director — Cochlear
Locations (3):
- Germany (2):
  - Deutsches HörZentrum Hannover der HNO-Klinik der MHH, Hanover, Lower Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Klinik für Hals, Nasen-, Ohrenheilkunde, Kopf und Halschirurgie, Kiel, Schleswig-Holstein
- Department of Otorhinolaryngology, Head and Neck Surgery, University Hospital, Zurich, Canton of Zurich, Switzerland